CLINICAL TRIAL: NCT04725110
Title: Phase II Trial of Direct Topical Lung T3 Treatment to Improve Outcome & Sequelae of COVID-19 ARDS - A Multi-Site, Randomized, Double-blinded, Placebo-Controlled Clinical Trial
Brief Title: Direct Topical Lung T3 Treatment to Improve Outcome & Sequelae of COVID-19 Acute Respiratory Distress Syndrome
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Duplicate record to NCT04115514
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PACCS-2020-23242
Record Dates: First submitted 2021-01-21; First posted 2021-01-26 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Covid19; SARS-CoV Infection; ARDS; ARDS, Human
MeSH Terms: conditions — COVID-19; Severe Acute Respiratory Syndrome; Respiratory Distress Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- T3 Intervention (Experimental): Participants in this arm will receive the experimental intervention.
  Interventions: Drug: Instilled T3
- Placebo Therapy (Placebo Comparator): Participants in this arm will receive placebo therapy.
  Interventions: Other: Placebo Therapy

INTERVENTIONS:
Drug: Instilled T3 — The first dose of T3 (50 micrograms in 10 mls volume BID) will be instilled by an investigator or under their direct supervision within 48 hours of obtaining consent after verifying that the patient is not too unstable to treat at that time. T3 doses will be given in 50 mcg doses twice daily for 4 days.
  Arms: T3 Intervention
Other: Placebo Therapy — A placebo therapy will be instilled into the lungs by the investigator or under their direct supervision within 48 hours of obtaining consent after verifying that the patient is not too unstable to treat at that time. Doses will be given twice daily for 4 days.
  Arms: Placebo Therapy

SUMMARY:
Acute treatment of COVID-ARDS with direct topical lung instilled T3 therapy for patients on mechanical ventilation.

DETAILED DESCRIPTION:
Post-hospitalization follow-up for 6 and 12-months of survival and end-organ dysfunction (lung, heart, kidney, neuropsychological), plus quality of life and return to work of those previously working

ELIGIBILITY:
Exclusion Criteria:

* Pregnancy

Inclusion Criteria:

* Diagnosis of SARS-CoV-2 with first positive test within 14 days, and,
* Diagnosis of ARDS by the Berlin Criteria (2012):

  1. Onset: < 7 days
  2. Chest x-ray: Bilateral Patchy Opacities, Infiltrates
  3. Mechanical Vent Support: PEEP or CPAP Support >= 5 cm H2O
  4. Pulmonary Edema: Not fully explained by cardiogenic etiology
  5. Hypoxia: PaO2/FIO2 Ratio < 300, or O2Sat/FIO2 Ratio < 315

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2030-10-15 (Estimated); Study Completion 2031-10-15 (Estimated)

PRIMARY OUTCOMES:
Change Extravascular Lung Water Index | 1 hour
  EVLWI is calculated as ml of extravascular lung water fluid reported by VolumeView system (Edwards Lifesciences) divided by patient's body weight in kg. EVLWI will be measured at baseline and 1 hour post T3 installation to calculate change in EVLWI. Lower EVLWI values indicate greater treatment efficacy.

SECONDARY OUTCOMES:
Length of ICU Stay | Baseline to ICU discharge up to 30 days
  Outcome is reported as the mean length of stay (in days) in the Intensive Care Unit (ICU) for participants in each arm.
Number of Ventilator-Free Days | 30 days
  Outcome is reported as the mean number of days participants in each arm did not require mechanical ventilation during an in-patient hospital admission.
30-day Survival | 30 days
  Outcome is reported as the number of participants in each arm who are alive 30-days post enrollment.
Creatinine Concentration | 4 days
  Outcome is reported as the number of participants in each arm with abnormally high plasma creatinine concentration (greater 1.21 milligrams per deciliter).
Glomerular Filtration Rate | 4 days
  Outcome is reported as the number of participants in each arm with impaired kidney function, defined as a glomerular filtration rate (GFR) less than 60 mL/min/1.73 m^2.
New York Heart Association (NYHA) Functional Classification | 30 days
  Outcome is reported as the number of participants in each arm who fall into each of 4 categories: 1 (no limitation in normal physical activity), 2 (mild symptoms only in normal activity), 3 (marked symptoms during daily activities, asymptomatic only at rest), and 4 (severe limitations, symptoms even at rest).

CONTACTS AND LOCATIONS:
Overall Officials: Timothy P Rich, MD, Principal Investigator — University of Minnesota; David Ingbar, MD, Study Chair — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States